CLINICAL TRIAL: NCT05699395
Title: Identification of Aortic Dissection Based on Pulse Oxygen and Ultrasound Doppler Waveforms
Brief Title: Quick Recognition of Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: QRAD2022
Record Dates: First submitted 2022-11-23; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-11

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aortic Dissection
  Interventions: Diagnostic Test: Non interventional
- Non Aortic Dissection
  Interventions: Diagnostic Test: Non interventional

INTERVENTIONS:
Diagnostic Test: Non interventional — No intervention

SUMMARY:
This is an observational study that establishes a cohort of patients with high risk chest pain who have been identified by CTA for aortic dissection. We then used this cohort to validate the accuracy of identifying aortic dissection based on extremity oximetry and Doppler waveforms.

ELIGIBILITY:
Inclusion Criteria:

* High risk chest pain with CTA

Exclusion Criteria:

* shock
* coma
* severe peripheral vascular diseases

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: High risk chest pain patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of aortic dissection | First 24-hours during emergency dapartment stay
  aortic dissection confirmed by CTA

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No